CLINICAL TRIAL: NCT00975468
Title: Prospective, Randomized Study of the Effects of Pressure-controlled vs. Volume-controlled Ventilation During One Lung Ventilation on Lung Injury After Thoracotomy
Brief Title: Pressure-Controlled vs Volume-Controlled Ventilation During One Lung Ventilation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial shortages due to lack of funderx
Sponsor: King Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCV vs. VCV during OLV; +966508491257
Record Dates: First submitted 2009-09-09; First posted 2009-09-11 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Thoracic Surgery
Keywords: pressure-controlled; volume-controlled; one lung; ventilation; lung injury; thoracotomy
MeSH Terms: conditions — Respiratory Aspiration; Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure-Controlled Ventilation (Active Comparator): The patients' lungs ventilation will be initiated with a peak airway pressure that provided a tidal volume of 8 ml.kg-1. R.R will be adjusted to achieve an arterial PaCO2 4.5-6 kPa and FiO2 will be increased to 1.0 during OLV.
  Interventions: Other: Pressure Controlled vs. Volume Controlled Ventilation during OLV
- Volume Controlled Ventilation (Placebo Comparator): The patients' lungs will ventilated with a tidal volume of 8 ml.kg-1. R.R will be adjusted to achieve an arterial PaCO2 4.5-6 kPa and FiO2 will be increased to 1.0 during OLV.
  Interventions: Other: Pressure Controlled vs. Volume Controlled Ventilation during OLV

INTERVENTIONS:
Other: Pressure Controlled vs. Volume Controlled Ventilation during OLV — Ventilation will be initiated with a tidal volume of 8 ml.kg-1 in Volume-controlled group and with a peak airway pressure that provided a tidal volume of 8 ml.kg-1 in pressure-controlled group. R.R will be adjusted to achieve an arterial PaCO2 4.5-6 kPa and FiO2 will be increased to 1.0 during OLV.

SUMMARY:
Compared with the information available in sepsis and trauma-associated ARDS, less is known about the cause and pattern of lung injury after thoracic surgery. Definition of lung injury in this context is difficult. Most now use the joint North American-European consensus conference definitions, but these are based only on gas exchange and radiology criteria. While gas exchange measures are reliable, thoracotomy inevitably causes radiological change and the interpretation of plain chest films becomes subjective. Definitions based on permeability and inflammatory changes would improve diagnosis, but are not routinely available in most units.

Pressure-controlled volume (PCV) may be useful to improve gas exchange and alveolar recruitment with associated lower airway pressures and shunt fraction during one-lung ventilation (OLV).

However, a recent prospective randomized study of the effects of PCV during OLV did not lead to improved oxygenation during OLV compared with VCV, but PCV did lead to lower peak airway pressures. To date, there are no reports of the effects of PCV versus VCV during OLV on the acute lung injury (ALI) after thoracotomy.

DETAILED DESCRIPTION:
Project Objectives:

We hypothesize that the use of PCV during OLV for thoracic surgery may improve the anti-inflammatory immunoregulation than VCV. It may attenuate the increases in proinflammatory cytokines, including interleukins (IL-8, IL-1, and IL-6) and TNF-α, and prevent suppression of the anti-inflammatory cytokine (IL-10) secretion.

The aims of the present study are:

Our research efforts will focus on identifying the effects of PCV vs.VCV during OLV for thoracotomy on the followings.

1. Intraoperative changes in the peak and plateau airway pressures and static and dynamic lung compliance.
2. Pulmonary function tests [vital capacity and FEV1] and arterial blood gases changes during the first 3 postoperative days.
3. The perioperative changes in serum levels of the proinflammatory cytokines, including IL-1, IL-6, IL8, and TNF-α and the anti-inflammatory cytokines IL-10,
4. The perioperative changes in BAL levels of the concentration of proteins, IL-1, IL-6, IL8, IL-10, and TNF-α.
5. The duration of postoperative ventilatory support, the time to extubation, the length of stay in post-anaesthesia care unit (PACU).
6. The incidence of the major complications (respiratory failure, cardiovascular events, bleeding, and renal dysfunction).

Project Design:

Study Design:

This prospective randomized placebo-controlled blinded study will be carried out from at the Cardiothoracic Surgery Unit - King Fahd University Hospital, after approval of the Institutional Ethical Committee.

Study Phases: The project comprised of five phases as follow:

• Phase I: Literature review collection and writing which will spend 2 months.

• Phase II: Pilot Study for 2 months to determine changes in the serum levels of cytokines to test the power of the study to define the proper sample size for both the VCV and PCV group during OLV.

• Phase III: A. Thoracic procedures using one-ling ventilation techniques: Arterial blood gases, chest X- ray, pulmonary function tests, liver function tests, CPK, samples collection [serum and BAL] and laboratory testing for cytokine changes.

B. Recording of the Clinical Outcome: included the times of ventilation, extubation, ICU and hospital stay, mortality and morbidity.

Sampling Site:

The study will be conducted in the OR suite and ICU at the King Fahd Hospital of the University - Alkhubar Study period: For 6 months. I. Patient Selection: patients aged 18-60 years (ASA physical status II-III) scheduled for elective open thoracic surgery using one lung ventilation for periods longer than 1.5 h will be allocated randomly to two groups by drawing of sequentially numbered sealed opaque envelopes that each contained a computer-generated randomization code. We will exclude the patients with decompensated cardiac (>New York Heart Association II), pulmonary diseases (VC or FEV1<50% of the predicted values), pulmonary hypertension (mean pulmonary artery pressure [MPAP] >30 mm Hg), and previous lobectomy or bilobectomy in the medical history, those treated with immune modulators (cytostatic drugs, corticosteroids and non-steroidal anti-inflammatory drugs, vaccination, blood products), within 3 months before surgery and with symptoms of an acute inflammatory process (clinically defined or abnormal data for C-reactive protein, leukocyte count, or body temperature).

II. Patient Groups and Study Protocol: Volume-controlled ventilation [VCV] group (n=according to the power of the study): patients' lungs will ventilated with a tidal volume of 8 ml.kg-1. Pressure-controlled ventilation [PCV] group (n=as before) patients' lungs ventilation will be initiated with a peak airway pressure that provided a tidal volume of 8 ml.kg-1. R.R will be adjusted to achieve an arterial PaCO2 4.5-6 kPa and FiO2 will be increased to 1.0 during OLV. All staff in the operating room, ICU and the ward will be unaware of the randomization code.

III. Anesthesia and Surgery: The patients will undergo combined thoracic epidural analgesia and general anesthesia using one lung ventilation technique for open thoracic surgical procedures through a standard posterolateral or an anterolateral muscle-sparing thoracotomy by the same consultants.

IV. The Investigators who will be involved with subsequent postoperative patient assessment will be blinded of the patient group.

V. Clinical Examination: included the intraoperative changes in airway pressures and lung compliances and the perioperative changes in pulmonary function tests [vital capacity and FEV1], the duration of postoperative ventilatory support, the time to extubation, the length of stay in PACU, the incidence of any major complications (respiratory failure, cardiovascular events, bleeding, and renal dysfunction).

VI. Blood Biochemistry: included the perioperative changes in arterial blood gases.

VII. Samples Collection and Analysis For the Inflammatory Mediators: The perioperative changes in serum levels of the concentration of the cytokines IL-1, IL-6, IL8, IL-10, and TNF-α, and the perioperative changes in BAL levels of the concentration of proteins, IL-1, IL-6, IL8, IL-10, and TNF-α.

1. . Type of samples: centrifuged stored aliquots of serum at -70°C and Supernatant frozen (at -80°C) broncho-alveolar lavage (BAL) aliquots.
2. . Laboratory Analysis:

   1. Cytokine determinations on the BAL fluid and plasma will be carried out using a solid-phase enzyme-linked immunosorbent assay method based on the quantitative immunometric sandwich enzyme immunoassay technique (Quantikine®; R&D Systems Ltd., Abingdon, UK).
   2. TNF-α immunoassay will be provided by Immunotech, France. Protein concentrations will be measured by an assay for the colorimetric detection and quantitation of total protein (Micro BCA TM Protein Assay Reagent Kit; Pierce, Rockford, IL).
   3. All samples of one patient will be analyzed in the same assay run.
   4. The samples will be measured in duplicates and the assays will be performed according to the manufacturer's instructions.
   5. The optical density of the samples will be determined by a microplate reader (Safire®; Tecan Ltd., Salzburg, Austria) and will be analyzed using the Safire microplate reader software by interpolation from standard curves. The sensitivities of the test kits are as follows: IL-1: 10 pg.mL-1, IL-6: 10 pg.mL-1, IL-8: 3.5 pg.mL-1, IL-10: 0.5 pg.mL-1, TNF : 5 pg.mL-1, protein: 0.5 µg.mL-1.

IV. Statistical Analysis: 2months Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS Inc., Chicago, IL). Data will be tested for normality using Kolmogorov-Smirnov test. An unpaired Student's t test will be used to compare the parametric values of the two groups; Mann-Whitney U test will be performed to compare the non-parametric values of the two groups. Serial changes in peri-operative data at the start of the treatment will be analyzed with repeated measures analysis of variance. PFTs variables and cytokine changes at different times within groups will be analysed with repeated measure analysis of variance (Anova test). Data will be expressed as mean (SD), number (%) or (median [range]). A value of P<0.05 will be considered to represent statistical significance.

V.Report Writing:2 months

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years (ASA physical status II-III) scheduled for elective open thoracic surgery using one lung ventilation for periods longer than 1.5 h

Exclusion Criteria:

We will exclude the patients with:

* decompensated cardiac (>New York Heart Association II)
* pulmonary diseases (VC or FEV1<50% of the predicted values)
* pulmonary hypertension (mean pulmonary artery pressure [MPAP] >30 mm Hg)
* previous lobectomy or bilobectomy in the medical history
* those treated with immune modulators (cytostatic drugs, corticosteroids and non-steroidal anti-inflammatory drugs, vaccination, blood products), within 3 months before surgery and with symptoms of an acute inflammatory process (clinically defined or abnormal data for C-reactive protein, leukocyte count, or body temperature)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Determine changes in the serum levels of cytokines | 4 months

SECONDARY OUTCOMES:
Arterial blood gases, chest X- ray, pulmonary function tests, samples collection [serum and BAL] and laboratory testing for cytokine changes, the times of ventilation, extubation, ICU and hospital stay, mortality and morbidity. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Regal, M.D, Study Director — King Faisal University
Locations (1):
- King Fahd Hospital of the University, Dammam, Eastern Province, Saudi Arabia